CLINICAL TRIAL: NCT01694576
Title: Adjuvant Chemotherapy or Not for NPC Patients Staged N2-3M0 After Concurrent Chemotherapy :a Phase Ⅱ Study
Brief Title: NPC Staged N2-3M0:Adjuvant Chemotherapy or Just Observation After Concurrent Chemoradiation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow patient enrollment
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Dr. Xia He, Director of the department of radiotherapy, Jiangsu Cancer Institute & Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC-N23-RCT; JSCC-RCT01 (Other: Department of Radiotherapy,Jiangsu Cancer Hospital)
Record Dates: First submitted 2012-09-17; First posted 2012-09-27 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma staged N2-3M0; Adjuvant chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Chemotherapy, Adjuvant; Paclitaxel; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant chemotherapy with paclitaxel and nedaplatin (Experimental): Patients will receive 3 cycles of adjuvant chemotherapy consisting of paclitaxel and platinum after concurrent chemoradiation
  Interventions: Drug: Adjuvant chemotherapy with paclitaxel and nedaplatin
- Observation (No Intervention): Patients will be followed up without adjuvant chemotherapy after concurrent chemoradiation

INTERVENTIONS:
Drug: Adjuvant chemotherapy with paclitaxel and nedaplatin — Patients receive 3 cycles of adjuvant chemotherapy consisting of paclitaxel and platinum after concurrent chemoradiation
  Other Names: Adjuvant chemotherapy
  Arms: Adjuvant chemotherapy with paclitaxel and nedaplatin

SUMMARY:
By this clinical trial, the investigators are trying to give an answer to such a question. Whether NPC patients staged N2-3M0 need adjuvant chemotherapy consisting of paclitaxel and platinum after concurrent chemoradiation?

DETAILED DESCRIPTION:
Recent research (Lancet Oncology 2012)shows that no survival benefits were achieved by adding adjuvant chemotherapy after concurrent chemoradiation in patients with locoregionally advanced NPC. But in patients with even high risk of distant metastasis(staged N2-3M0),is adjuvant chemotherapy necessary?

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed untreated NPC patients staged N2-3M0
2. age: 18y - 65y
3. with MRI examinations
4. ECOG≤2
5. with written consent

Exclusion Criteria:

1. without a second cancer
2. pregnancy
3. with other severe diseases(blood,liver ,kidney or heart diseases)
4. could not staged properly
5. without written consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
treatment toxicity based on a CTCAE3.0 grading system | 6 months

SECONDARY OUTCOMES:
progress free survival | 24 months

OTHER OUTCOMES:
distant metastasis free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Xia He, M.D. and PhD, Principal Investigator — Department of Radiotherapy,Jiangsu Cancer Hospital
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China